CLINICAL TRIAL: NCT06507241
Title: Clinical and Instrumental Assessment of Meniscal ROOT Tears Treated Through Suture to the Posterior Cruciate Ligament
Acronym: ROOT-PCL
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Full Professor Medicine and Surgery, University of Bologna, Istituto Ortopedico Rizzoli
Other Study IDs: ROOT-PCL
Record Dates: First submitted 2024-07-04; First posted 2024-07-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Meniscus Tear; Meniscus Lesion; Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The menisci are crucial for knee stability and functionality. Composed of fibrocartilaginous structure, they have an anatomical and biomechanical arrangement that makes them essential for load transmission and the prevention of osteoarthritis. Meniscal root lesions, known as "ROOT tears," compromise their protective function on the cartilage, leading to increased contact pressures between the tibia and femur and, over time, the development of osteoarthritis. Early diagnosis of these lesions is difficult and often the first detection is incidental. The subsequent challenges are significant due to a lack of pre-operative planning. A possible solution is a surgical technique involving arthroscopic suture of the posterior meniscal root along with the posterior cruciate ligament. This procedure does not require pre-operative planning and is applicable even in cases of incidental diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 50 years at the time of surgery;
2. Male and female gender;
3. Patients undergoing surgical treatment for at least one year for "ROOT" type meniscal lesions using arthroscopic suturing to the posterior cruciate ligament;
4. Pre-operative MRI performed.

Exclusion Criteria:

1. Patients no longer reachable;
2. Patients who refuse consent to the study;
3. Previous meniscectomy before surgery;
4. Previous ligament injuries before surgery;
5. New traumatic injuries after surgery;
6. Advanced knee osteoarthritis (Outerbridge grade III-IV) at the time of surgery;
7. Severe knee malalignment (> 5°) at the time of surgery;
8. Severe obesity (BMI > 35);
9. Lower limb conditions preventing full weight-bearing during evaluation;
10. Infection or hematological/rheumatic conditions at the time of evaluation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be recruited among all subjects with "ROOT" type meniscal lesions treated surgically with arthroscopic suturing to the posterior cruciate ligament (ROOT-PCL) from 1/1/2021 to 31/12/2025 at the Rizzoli Orthopedic Institute.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
RMN | 24 months after surgery
  The 3 Tesla MRI is the diagnostic test of choice used in common clinical practice to evaluate the healing of these lesions at 1 and 2 years of follow-up. The measured parameter is meniscal extrusion. The measurement is taken in millimeters at the coronal sections visualizing the medial collateral ligament, from the capsular margin of the body to the outer profile of the tibial plateau. The "ghost sign" and tibial plateau edema will also be looked for. The main limitation of MRI is related to the fact that it is performed non-weight-bearing, with the patient in a supine position.

SECONDARY OUTCOMES:
Weight-bearing ultrasound | 24 months after surgery
  Weight-bearing ultrasound is a method not commonly used in clinical practice but extremely useful in evaluating meniscal extrusion under conditions close to physiology. The measurement is performed in a static position with the patient standing upright with full weight-bearing. Once again, meniscal extrusion is measured in millimeters in the coronal sections visualizing the medial collateral ligament, from the capsular margin of the body to the outer profile of the tibial plateau. The strength of this method lies in its ability to replicate the biomechanical stress phenomena affecting the menisci during common daily activities, with the potential to detect lesions that would otherwise remain silent in a non-weight-bearing MRI.
Physical examination | 24 months after surgery
  A comprehensive assessment will include palpation to identify classic tender points related to meniscal pathology at the anterior, middle, and posterior joint lines. The presence of pain and the patient's overall health status will then be noted.
International Knee Documentation Committee (IKDC) | 24 months after surgery
  The IKDC form evaluates knee function subjectively across three domains: Symptoms (including pain, stiffness, swelling, and locking), Sports and daily activities, and Current knee function compared to before injury. It consists of 10 questions focusing on symptoms, sports participation, daily activity difficulties, and current knee function. Scores range from 0 to 100, with higher scores indicating better knee health: excellent (80-100), good (60-80), fair (30-60), and poor (0-30).
Lysholm Knee Score | 24 months after surgery
  It's a validated measurement scale that assesses knee functionality through 8 items, allowing to establish the knee's condition in relation to the functional demands of daily life activities. This assessment tool is used to evaluate surgical outcomes in patients who have undergone knee ligamentous or meniscal injuries. The final score is derived from the sum of various scores obtained across different items, ranging from 0 to 100. Scores are categorized into subgroups: Excellent (95-100); Good (84-94); Fair (65-83); Poor (<64).
VAS (Visual Analog Scale) | 24 months after surgery
  It is a quantitative one-dimensional numerical scale for pain assessment with 10 points; the scale requires the patient to select the number that best describes the intensity of their pain from 0 to 10 at that specific moment. 0 indicates no pain, while 10 indicates the worst possible pain.
Tegner Score | 24 months after surgery
  It allows estimation of the level of motor activity of a subject with a score ranging from 0 to 10, where 0 represents 'disability' and 10 represents 'participation in competitive sports such as national or international-level soccer'. This score is widely used to define the level of motor activity in patients with knee disorders. In the study, the Tegner Score will be completed directly by the investigator through an interview with the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy